CLINICAL TRIAL: NCT05710575
Title: Role of Probiotic Use in Outcomes of Premature Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Collaborators: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Komal Khadim Hussain, principal investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB/2022/920/SIMS
Record Dates: First submitted 2023-01-13; First posted 2023-02-02 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Necrotizing Enterocolitis of Newborn
Keywords: probiotic; premature birth
MeSH Terms: conditions — Premature Birth | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomization will be carried out in blocks of 10, and the list of random numbers will be generated by the subprogram Epitable from Epi-Info 6.04 (Centers for Disease Control and Prevention, Atlanta, GA). Two trained external personnel from the NICU will be responsible for obtaining this list and for randomly assigning the infants to the probiotics and control groups. A sealed envelope with the identification number in ascending order, containing information about which group they belonged to, will be provided for each infant and will be sent to the hospital's nutritional center. Three previously trained research assistants, who will not be a part of the neonatal team, will interview the mothers, recruit the infants, and they will also be responsible for sending the envelopes to the nutritional unit.
Who Masked: Participant
Masking Description: Randomization will be carried out in blocks of 10, and the list of random numbers will be generated by the subprogram Epitable from Epi-Info 6.04 (Centers for Disease Control and Prevention, Atlanta, GA). Two trained external personnel from the NICU will be responsible for obtaining this list and for randomly assigning the infants to the probiotics and control groups. A sealed envelope with the identification number in ascending order, containing information about which group they belonged to, will be provided for each infant and will be sent to the hospital's nutritional center. Three previously trained research assistants, who will not be a part of the neonatal team, will interview the mothers, recruit the infants, and they will also be responsible for sending the envelopes to the nutritional unit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- probiotic group (Experimental): Probiotic or placebo administration will be started from the first feed of the infants. Infants in the probiotic group will receive five drops of oil-based suspension containing 1×108 colony-forming units of L reuteri (DSM 17938 Biogaia AB, Stockholm, Sweden) once a day, until death or discharge from the hospital. For infants on oral feeds, after suctioning oral secretions, five drops will be placed in the posterior oropharynx of the infants. For infants without per oral feeds, five drops will be administered through a gastric tube followed by a flash of 0.5 mL of sterile water. For the infants in the placebo group, five drops from an identical vial containing only oil base will be administered following the same protocol as the probiotic group.
  Interventions: Biological: probiotic
- placebo group (Experimental): Probiotic or placebo administration will be started from the first feed of the infants. Infants in the probiotic group will receive five drops of oil-based suspension containing 1×108 colony-forming units of L reuteri (DSM 17938 Biogaia AB, Stockholm, Sweden) once a day, until death or discharge from the hospital. For infants on oral feeds, after suctioning oral secretions, five drops will be placed in the posterior oropharynx of the infants. For infants without per oral feeds, five drops will be administered through a gastric tube followed by a flash of 0.5 mL of sterile water. For the infants in the placebo group, five drops from an identical vial containing only oil base will be administered following the same protocol as the probiotic group.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: probiotic — Probiotic or placebo administration will be started from the first feed of the infants. Infants in the probiotic group will receive five drops of oil-based suspension containing 1×108 colony-forming units of L reuteri (DSM 17938 Biogaia AB, Stockholm, Sweden) once a day, until death or discharge from the hospital. For infants on oral feeds, after suctioning oral secretions, five drops will be placed in the posterior oropharynx of the infants. For infants without per oral feeds, five drops will be administered through a gastric tube followed by a flash of 0.5 mL of sterile water. For the infants in the placebo group, five drops from an identical vial containing only oil base will be administered following the same protocol as the probiotic group.
  Arms: probiotic group
Other: placebo — Probiotic or placebo administration will be started from the first feed of the infants. Infants in the probiotic group will receive five drops of oil-based suspension containing 1×108 colony-forming units of L reuteri (DSM 17938 Biogaia AB, Stockholm, Sweden) once a day, until death or discharge from the hospital. For infants on oral feeds, after suctioning oral secretions, five drops will be placed in the posterior oropharynx of the infants. For infants without per oral feeds, five drops will be administered through a gastric tube followed by a flash of 0.5 mL of sterile water. For the infants in the placebo group, five drops from an identical vial containing only oil base will be administered following the same protocol as the probiotic group.
  Arms: placebo group

SUMMARY:
Project Summary:

The prevalence of preterm birth ranges from 5% to 18% across 184 countries, and an estimated 15 million infants are born preterm globally. These infants with an immature immune system and gastrointestinal tract are at risk of complications of premature birth, which is the leading cause of neonatal death. According to researcher hypothesis for this study, there is role of probiotics in promoting food tolerance and reducing the incidence and severity of Necrotizing Enterocolitis (NEC) and death related to NEC in pre-term VLBW infants. In the current study, we will examine the effects of probiotics in premature infants and figure out the optimal intervention through randomized controlled trial (RCT).

A prospective, masked, randomized single blinded controlled trial will be conducted in the neonatal intensive care unit (NICU) of Services Hospital Lahore. In this trial the treatment group will receive the probiotics during their first month of life, and the control group will receive no treatment. Primary outcome will be the incidence of death or NEC (≥ stage 2). Death is included as a primary outcome because it is a competing variable of NEC. The x2 test will be used to analyze the categorical data, along with Fisher's exact test when applicable. The Student's t test will be used for continuous data. A logistic regression model will be used to analyze the treatment effects on the primary and secondary outcome variables (death, NEC, and sepsis). Values will be expressed for mean and standard deviation. Statistical significance is set at P-value of 0.05.

The objective of this study is to confirm the evidence and to get the more reliable and authentic results regarding the more effective treatment of NEC in preterm neonates. In this way, the researcher shall be able to improve the outcome of premature births and to reduce the complications by increasing the cure rate. Similarly, it will help the researcher to improve knowledge for better management of NEC in neonates.

DETAILED DESCRIPTION:
Despite improvement in antenatal services, preterm births have remained a common but serious problem. In recent years because of environmental factors and increase rate of in vitro fertilization, the prevalence of preterm birth ranges from 5% to 18% across 184 countries, and globally, the number of infants with preterm birth is around 15 million. . These infants, with immature immune system and gastrointestinal tract, are at risk of complications of premature birth, which is a leading cause of neonatal death .

Recent studies suggest that the composition of infants' gut micro biota is affected by birth weight and gestational age. Altered gut micro biota has proven to be an important factor putting infants at high risk of developing necrotizing enterocolitis (NEC) and sepsis, which may lead to death and lifelong physical impairment. It is evident that early probiotic supplementation may benefit premature infants by improving their gastrointestinal tolerance against potential pathogens and regulating the altered gut micro biota to resemble that of a term healthy infant.

Probiotic with or without prebiotic supplementation is a practicable method among nutrition interventions and may support gut micro biota colonization growth, and long-term neurologic development in premature infants. Probiotic supplements in formula may regulate the stability and composition of premature infants' gut microbiota. Recent studies and meta-analyses suggest that probiotic intervention has some positive effects on premature infants, especially in reducing the mortality and morbidity of NEC and sepsis. Deshpande et al. showed that probiotics could reduce the risk of late-onset sepsis and NEC when Bifidobacterium or Lactobacillus was part of the supplementation through a subgroup analysis in pairwise meta-analysis, but the result was restricted to low- and middle-income countries. However, previous pairwise meta-analysis only focused on efficacy but could not find the most effective intervention method. It is suggested that there are different effects when different strains or combinations are used.

As numerous strains and preparations, including multi strains without given reasons, have been used in relevant trials, probiotic usage in infants needs to be regulated by more evidence. Previously published network meta-analyses in which authors compare the effect of different strains also have several shortcomings in their methodology or design. Thus, the authors of these studies did not point out which strain is an optimum option for infants' health and failed to provide powerful evidence for clinical use of probiotics. In the current study, the researchers will examine the effect of probiotics in premature infants and will figured out the optimal intervention through randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Premature infants with gestational age of more than 28 weeks and less than 36 weeks
* Birth weight of 1000 - 2500 grams
* Admitted to the neonatal intensive care unit (NICU) of Pediatric Medicine Unit II, Services hospital Lahore
* With intestinal feeding.

Exclusion Criteria:

* Infants with major congenital malformations (including congenital heart disease, gastrointestinal obstruction, gastroschisis, etc.)
* Congenital metabolic errors hypoxic ischemic encephalopathy (HIE) of grade two or more according to Sarnat scoring system (Gordon et al., 2020)
* Death in the first 72 hours of life
* Newborns of addicted mothers
* Postpartum age more than two weeks
* Parental unacceptance

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
number of participants who develop necrotizing enterocolitis | 1 month
  necrotizing enterocolitis will be stage according to bell's staging
number of participants with prolonged hospital stay | 1 month
  length of hospital stay from day of admission to day of discharge according to medical records

SECONDARY OUTCOMES:
number of participants with culture proven sepsis | 1 month
  culture proven sepsis in premature infants after taking probiotics
number of participants with feeding intolerance | 1 month
  premature infants unable to take feed and at what time infants achieve fll enteral feed

CONTACTS AND LOCATIONS:
Overall Officials: komal khadim hussain, MBBS, Principal Investigator — Services Institute of Medical Sciences, Pakistan; dr azhar farooq, MBBS,FCPS, Study Chair — Services Institute of Medical Sciences, Pakistan
Locations (1):
- services hospital Pakistan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No